CLINICAL TRIAL: NCT06262607
Title: A Randomized, Double-blind, Vehicle-controlled, Multicenter, Parallel-Design, Phase 2 Study to Assess the Efficacy and Safety of CLE-400 Topical Gel for the Treatment of Chronic Pruritus in Adult Subjects With Notalgia Paresthetica
Brief Title: A Study of CLE-400 (Topical Gel) for the Treatment of Chronic Pruritus in Adult Subjects With Notalgia Paresthetica
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clexio Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLE400-NP-201
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pruritus in Adult Subjects With Notalgia Paresthetica (NP)

STUDY DESIGN:
Intervention Model Description: 54 subjects, 2 arms, parallel
Who Masked: Participant, Investigator
Masking Description: double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CLE-400 (Detomidine topical gel) (Experimental): Topical CLE-400 gel 0.28% once daily
  Interventions: Drug: CLE-400
- Vehicle (Placebo Comparator): Topical vehicle gel once daily
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: CLE-400 — Topical CLE400 gel 0.28% administered once daily
  Arms: CLE-400 (Detomidine topical gel)
Drug: Vehicle — Topical vehicle gel administered once daily
  Arms: Vehicle

SUMMARY:
This is a Phase 2, randomized, double-blind, vehicle-controlled study to assess the efficacy and safety of CLE-400 topical gel for the treatment of chronic pruritus in adult subjects with Notalgia Paresthetica (NP).

DETAILED DESCRIPTION:
Study to assess the efficacy and safety of CLE-400 topical gel applied once daily for the treatment of moderate-severe chronic pruritus in adult subjects with NP. The study comprises a screening phase of up to 37 days, including a 7-day run-in period, a 4-week double-blind treatment period, and a 2-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed diagnosis of Notalgia Paresthetica.
* Subject has a history of chronic pruritus (itch) due to Notalgia Paresthetica.
* Subject has moderate to severe pruritus.
* Subject is able and competent to read and sign the informed consent form (ICF).

Exclusion Criteria:

* Subject has chronic pruritus that is related to a condition other than Notalgia Paresthetica.
* Subject with known or suspected history of a clinically significant systemic disease, unstable medical disorders, life-threatening disease, including physical/laboratory/ECG/vital signs abnormality that would put the subject at undue risk or interfere with interpretation of study results
* Subject is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Clinical site 11, Bryant, Arkansas
  - Clinical Site 21, Fremont, California
  - Clinical site 01, Coral Gables, Florida
  - Clinical Site 13, Margate, Florida
  - Clinical Site 10, North Miami Beach, Florida
  - Clinical Site 02, Indianapolis, Indiana
  - Clinical Site 23, Methuen, Massachusetts
  - Clinical Site 20, Portsmouth, New Hampshire
  - Clinical Site 15, New York, New York
  - Clinical site 03, High Point, North Carolina
  - Clinical Site 09, Dublin, Ohio
  - Clinical site 16, Houston, Texas
  - Clinical Site 06, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CLE-400 (Detomidine Topical Gel) | Vehicle
Started | 28 | 31
Completed | 26 | 30
Not Completed | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CLE-400 (Detomidine Topical Gel) | Vehicle | Total
Number analyzed (Participants) | 28 | 31 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 20 | 38
  >=65 years | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.82 (8.2) | 60.48 (10.5) | 61.12 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 17 | 20 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 27 | 29 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 31 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Weekly Mean of the Daily 24-hour Worst Itch-Numeric Rating Scale (WI-NRS) Score at Week 4.
Description: The WI-NRS is a tool used to assess the intensity of the most severe (worst) pruritus (itch), as experienced by the subject, in the last 24 hours. WI-NRS scale score ranges from 0 to 10, with 0 indicating no itch and 10 indicating the worst itch imaginable.
Time Frame: Baseline, Week 4 (28 days).
Population: The FAS is a subset of the ITT analysis set and will include all randomized subjects who received at least 1 dose of study treatment and have both baseline and at least one post-baseline weekly mean WI-NRS evaluation. In this analysis set, treatment is assigned based on the treatment to which subjects were randomized, regardless of which treatment they actually received. The FAS serves as the principal analysis set for efficacy inference.
Measure: Least Squares Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | CLE-400 (Detomidine Topical Gel) | Vehicle
Number analyzed (Participants) | 28 | 31
percentage of change from baseline | -44.37 (5.75) | -50.37 (5.43)
Statistical Analysis 1: Comparison: CLE-400 (Detomidine Topical Gel) vs Vehicle; Test type: Superiority; p = 0.4422, Mixed Models Repeated Measures (MMRM); Least square (LS) mean difference = 6.0, 95% CI 2-sided [-9.54 to 21.53], Standard Error of Mean 7.74

ADVERSE EVENTS:
Time Frame: 6 weeks after participant received first dose
Arm/Group | CLE-400 (Detomidine Topical Gel) | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/31
Other Adverse Events (participants affected / at risk) | 8/28 | 5/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLE-400 (Detomidine Topical Gel) (N=28) | Vehicle (N=31)
Application site paraesthesia (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Xerosis (General disorders) | 0 (0) | 1 (1)
Pyuria (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or 18 months after completion of the Study, whichever occurs first, Institution may itself publish the results of its data from the Study. Institution and Principal Investigator shall provide Sponsor with an advance copy of any proposed publication or oral presentation at least 60 days prior to the planned date of submission or presentation and Sponsor shall have 60 days to review the proposed publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT06262607/Prot_SAP_000.pdf